CLINICAL TRIAL: NCT00775619
Title: An Open Label, Balanced, Randomised, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover Bioavailability Study on Carvedilol Formulations Comparing Carvedilol 12.5 mg Tablets of Ranbaxy Laboratories With Coreg® 12.5 mg Tablets of Glaxosmithkline in Healthy, Adult, Human Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Carvedilol 12.5mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 023/CARVE-12.5/03
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence Carvedilol 12.5 mg tablets fed conditions
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Coreg® 12.5 mg tablets
  Interventions: Drug: Carvedilol 12.5 mg tablets
- 1 (Experimental): Carvedilol 12.5 mg tablets
  Interventions: Drug: Carvedilol 12.5 mg tablets

INTERVENTIONS:
Drug: Carvedilol 12.5 mg tablets — bioequivalence Carvedilol 12.5 mg tablets fed conditions

SUMMARY:
The objective of this study was to compare the single-dose oral bioavailability of Carvedilol 12.5 mg tablets of Ranbaxy Laboratories with Coreg 12.5 mg tablets of Glaxosmithkline in healthy, adult, human subjects under fed conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover, bioavailability study on carvedilol formulation comparing carvedilol 12.5mg of Ohm Laboratories, Inc. (a subsidiary of Ranbaxy pharmaceuticals Inc, USA) with Coreg® 12.5mg tablet (containing carvedilol 12.5 mg) of GlaxoSmithKline, USA in healthy, adult, male, human subjects under fed condition.

Forty healthy, adult, human subjects who met the inclusion and exclusion criteria as described in the protocol were enrolled in the study. Thirty-nine subjects completed both the periods of the study

ELIGIBILITY:
Inclusion Criteria:

* Be in the' age range of 18-45 years.
* Be neither overweight nor underweight for his/her height as per the Life Insurance Corporation of lndia height/weight chart for non-medical cases.
* Have voluntarily given written informed consent to participate in this study.
* Be of normal health as determined by medical history and physical examination of the subjects performed within :1.4 days prior to the commencement of the study.

If female and:

* Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device ([UD), or abstinence; or Is postmenopausal for at least 1 year; or
* Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* History of allergy to 13-adrenoceptor antagonists especially carvedilol.
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Presence of disease markers of HIV 1 and 2, Hepatitis B and C viruses or syphilis infection.
* Female volunteers demonstrating a positive pregnancy test.
* Female volunteers who are currently breastfeeding.
* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.

Positive for urinary screen testing of drugs of abuse (opiates And cannabinoids)

* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray.
* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes, glaucoma, bronchial asthma, fainting or syncope.
* History of any psychiatric illness which may impair the ability to provide written informed consent.
* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on Habitual basis of more than 2 units of alcoholic beverages per day (1 Unit equivalent to half pint of beer or ! glass of wine or I measure of spirit) or have difficulty_ in abstaininq for the duration of each study period.
* Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
* A haemoglobin concentration of less than 7 % of lower limit of reference range e.g. 13 gm % for reference range of 1448 gm at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html